CLINICAL TRIAL: NCT01955603
Title: A Randomised, Placebo-controlled, Double-blind Within Cohort, Dose Escalation, Multiple-dose Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0215-0384 Administered Subcutaneously to Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC0215-0384 Administered to Subjects With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8210-3927; 2012-003969-18 (EudraCT Number); U1111-1133-7983 (Other: WHO)
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid | interventions — NNC0215-0384

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose level 1 (Experimental)
  Interventions: Drug: NNC0215-0384; Drug: placebo
- Dose level 2 (Experimental)
  Interventions: Drug: NNC0215-0384; Drug: placebo
- Dose level 3 (Experimental)
  Interventions: Drug: NNC0215-0384; Drug: placebo

INTERVENTIONS:
Drug: NNC0215-0384 — A total of seven once-weekly doses of NNC0215-0384 or placebo will be administered subcutaneously (s.c., under the skin) at one of three ascending dose levels. Each cohort will consist of eight subjects randomised to either active (6 subjects) or placebo (2 subjects) treatment. Each subject will participate in one cohort only. Dose-escalation to the next dose level will be initiated when the safety data has been evaluated and if considered safe.
Drug: placebo — Placebo administered corresponding to NNC0215-0384 treatment

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability, pharmacokinetics (exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of NNC0215-0384 administered to subjects with moderate to severe rheumatoid arthritis (RA) concomitantly treated with methotrexate (MTX).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age between 18 and 75 years (both years inclusive), for Russia only: Age between 18-65 years (both years inclusive)
* Moderate to severe RA, confirmed by a Disease Activity Score based on 28 joints and C-reactive protein (DAS28 (CRP)) equal to or above 4.5 and a minimum of five tender and five swollen joints based on a 28 joint count (a joint can score as both tender and swollen)
* MTX (10-25 mg/week both inclusive) for at least 16 weeks, with an unchanged dose for at least 6 weeks prior to screening and until randomisation
* Females who are not of child-bearing potential must have been post-menopausal for at least 1 year confirmed by follicle-stimulating hormone (FSH) equal to or above 26.7 U/L or be surgically sterile

Exclusion Criteria:

* Past or current inflammatory joint disease other than RA (e.g. gout [crystal proven], psoriatic arthritis, juvenile idiopathic arthritis, reactive arthritis or Lyme disease
* Any active or ongoing chronic infectious disease (e.g. chronic osteomyelitis, chronic pyelonephritis) within 4 weeks prior to randomisation
* Clinically significant cardiac or cardiovascular disease
* Past or current malignancy
* Evaluation of tuberculosis screening indicative of latent or active tuberculosis (TB)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From first dosing until 19 weeks after first dosing

SECONDARY OUTCOMES:
Concentration of NNC0215-0384 in serum | 7 days after each dose
Concentration of NNC0215-0384 in serum | 3 days after first and last dose
Duration of full and duration of detectable levels of C5a receptor (C5aR) occupancy by NNC0215-0384 on neutrophils from baseline | From week 0 until 19 weeks after first dosing
Change in health assessment questionnaire - disability index (HAQ-DI) from baseline | Week 0, week 7 first dosing
Incidence and characterisation of antibodies directed against NNC0215-0384 and, if present, their in vitro neutralising activity | From first dosing until 19 weeks after first dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (4):
- Berlin, Germany
- Budapest, Hungary
- Krakow, Poland
- Moscow, Russia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com